CLINICAL TRIAL: NCT04394520
Title: A Randomized Controlled Trial of Varying Consent Language and Mode to Improve Interactive Voice Response (IVR) Survey Performance in Colombia and Uganda
Brief Title: Use of Consent Language and Mode to Improve Interactive Voice Response Survey in Colombia and Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other); Makerere University (Other); Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-6.1
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; consent
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of five introduction and consent combinations: 1) standard introduction and standard consent mode (active opt-in and active opt-out); 2) modified introduction language and standard consent mode; 3) modified introduction language and active opt-in consent; 4) modified introduction language and active opt-out consent; or 5) modified introduction language and passive opt-in consent. This randomization will occur at the beginning of the survey.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): No change will be made to the introduction content or the consent mode (active opt-in and active opt-out) from other related trials
- Modified Intro, Standard Consent (Experimental): Modified introductory language will be used, but the consent structure (active opt-in and active opt-out) will remain the same.
  Interventions: Other: Modified Introduction
- Modified Intro, Active Opt-in (Experimental): Modified introductory language will be used, and the consent mode will be changed to active opt-in only.
  Interventions: Other: Modified Introduction; Other: Active Opt-in
- Modified Intro, Active Opt-out (Experimental): Modified introductory language will be used, and the consent mode will be changed to active opt-out only.
  Interventions: Other: Modified Introduction; Other: Active Opt-out
- Modified Intro, Passive Opt-in (Experimental): Modified introductory language will be used, and the consent mode will be changed to passive opt-in only.
  Interventions: Other: Modified Introduction; Other: Passive Opt-in

INTERVENTIONS:
Other: Modified Introduction — A variation in the introductory content to motivate participants to complete the survey. Participants will be presented with modified introductory language based on the findings from local focus groups and key informant interviews.
  Arms: Modified Intro, Active Opt-in; Modified Intro, Active Opt-out; Modified Intro, Passive Opt-in; Modified Intro, Standard Consent
Other: Active Opt-in — A variation in the consent mode to motivate participants to complete the survey. Participants will be given the choice to actively opt-in to the survey, if they do not respond, the survey will terminate.
  Arms: Modified Intro, Active Opt-in
Other: Active Opt-out — A variation in the consent mode to motivate participants to complete the survey. Participants will be given the choice to actively opt-out to the survey, if they do not respond, the survey will continue.
  Arms: Modified Intro, Active Opt-out
Other: Passive Opt-in — A variation in the consent mode to motivate participants to complete the survey. Participants will be given the choice to passively opt-in to the survey, if they do not hang-up, the survey will continue.
  Arms: Modified Intro, Passive Opt-in

SUMMARY:
This study evaluates the effect of one new form of introduction language and three new modes of providing consent on interactive voice response (IVR) survey cooperation, response, refusal and contact rates, as compared to control group, in Colombia and Uganda.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technique, RDD participants will be randomized to one of five introduction and consent combinations and then have them complete noncommunicable disease risk factor survey with an additional module regarding their understanding of the survey and of its voluntariness. This mobile phone survey will be sent as an interactive voice response (IVR). In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. If you are male, press 1; If you are female, press 2). This study will be conducted in both Colombia and Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Colombia, conversant in the Spanish language. In Uganda, conversant in Luo, Luganda, Runyakitara or English languages.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3786 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, the number of complete interviews divided by the number of complete interviews, partial interviews, refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, the number of complete and partial interviews divided by the number of complete interviews, partial interviews, refusals, breakoffs and the estimated eligible proportion of unknowns.

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, the number of refusals and breakoffs divided by the number of complete interviews, partial interviews, refusals, breakoffs and the estimated eligible proportion of unknowns.
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, the number of complete and partial interviews, refusals and breakoffs divided by the number of complete interviews, partial interviews, refusals, breakoffs and the estimated eligible proportion of unknowns.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W. Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Instituto de Salud Publica Pontificia Universidad Javeriana, Bogotá, D.C., Colombia
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722